CLINICAL TRIAL: NCT01205477
Title: Phase 2 Double-blinded, Placebo-controlled, Clinical Trial for Safety and Efficacy of Methylprednisolone Infiltration in Anserine Bursitis Treatment
Brief Title: Safety and Efficacy of Methylprednisolone Infiltration in Anserine Bursitis Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: David Vega Morales, Departamento de Reumatología, Hospital Universitario "José Eleuterio González" de la Universidad Autónoma de Nuevo León
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RE09-009
Record Dates: First submitted 2010-07-28; First posted 2010-09-20 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2009-06

CONDITIONS: Bursitis
Keywords: Anserine bursitis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisolone (Experimental): Infiltration of 40 mg of methylprednisolone acetate plus 1 mL of xylocaine
  Interventions: Drug: EXPERIMENTAL
- Placebo (Placebo Comparator): Infiltration of 1 mL of xylocaine
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: EXPERIMENTAL — Infiltration of 40 mg of methylprednisolone acetate plus 1 mL of xylocaine and Diclofenac sodium 100 mg PO QD for 10 days
  Other Names: DEPOMEDROL
  Arms: Methylprednisolone
Drug: PLACEBO — Infiltration of 1 mL of xylocaine and Diclofenac sodium 100 mg PO QD for 10 days
  Arms: Placebo

SUMMARY:
To investigate the safety and efficacy of methylprednisolone infiltration in anserine bursitis treatment

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of anserine bursitis

Exclusion Criteria:

* Intraarticular pathology that reflects pain in the medial part of the knee

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
WOMAC score | 4 weeks
  The WOMAC (Westren Ontario and McMaster Universities) index is used to assess patients with osteoarthritis of the hip or knee using 24 parameters. It can be used to monitor the course of the disease or to determine the effectiveness of anti-rheumatic medications.
  Pain, Stiffness and Physical functionVisual analogue scale (VAS) may be used ranging from 0 to 10.

SECONDARY OUTCOMES:
VAS satisfaction | 4 weeks
  Visual Analoge Scale for satisfaction
Improvement | 4 weeks
  Percentage of improvement
SAFETY | 4 weeks
  Pain at infiltration site, ecchymosis, bleeding, paresthesias, skin infection, anaphilaxy, vasovagal reaction

CONTACTS AND LOCATIONS:
Overall Officials: Mario Alberto Garza Elizondo, MD, Study Director — Universidad Autónoma de Nuevo León
Locations (1):
- Hospital Universitario "José Eleuterio González", Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Alvarez-Nemegyei J, Canoso JJ. Evidence-Based Soft Tissue Rheumatology IV: Anserine Bursitis. J Clin Rheumatol. 2004 Aug;10(4):205-6. doi: 10.1097/01.rhu.0000135561.41660.b0. PMID 17043509
- [Background] Calvo-Alén J, Rua-Figueroa I, Erausquin C. Anserine bursitis treatment: local corticoesteroid injction against NSAID: a prospective study [Spanish]. Rev Esp Reumatol. 1993;20:13-15.